CLINICAL TRIAL: NCT00356668
Title: Observational, Cross-over Study of the Positive Distending Pressure Generated by Humidified High Flow Nasal Cannula as Compared to Nasal Continuous Positive Airway Pressure
Brief Title: Humidified High Flow Nasal Cannula as Compared to Nasal Continuous Positive Airway Pressure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0606-051
Record Dates: First submitted 2006-07-24; First posted 2006-07-26 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Respiratory Distress Syndrome; Cronic Lung Disease
Keywords: HFNC; NCPAP; nasal continuous positive airway pressure; humidified high flow nasal cannula; esophageal pressure; gas flow
MeSH Terms: conditions — Respiratory Distress Syndrome

INTERVENTIONS:
Device: High Flow Nasal Cannula — 30 minute blocks on varying flows of high flow nasal cannula

SUMMARY:
The specific aims of this study are to evaluate the amount of high flow nasal cannula (HFNC) gas flow required to generate an equivalent positive distending pressure as that provided by nasal continuous positive airway pressure (NCPAP) of 6 cm H2O, assess the relationships between positive distending pressure, gas flow, oxygen requirement, and patient weight, and lastly, develop an appropriate protocol to be used in the NICU for transitioning patients from NCPAP to an equivalent amount of HFNC.

DETAILED DESCRIPTION:
In the face of exogenous surfactant and use of antenatal steroids, respiratory distress syndrome (RDS) remains a leading cause of morbidity and mortality in premature infants. RDS is the result of a series of complex, interrelated events, including atelectasis, ventilation-perfusion mismatching, and lung inflammation/injury (1). The cascade of events which typifies RDS and its long-term counterpart, chronic lung disease (CLD), is rooted in the intrinsic deficits of the premature lung as well as exacerbated by mechanical ventilation, a mainstay of therapy. For this reason, scientists and clinicians alike continue to search for treatment modalities which will not only treat RDS but also decrease the incidence of chronic lung disease.

The use of non-invasive ventilatory strategies, such as nasal continuous positive airway pressure (NCPAP), in the treatment of RDS is thought to provide positive distending pressure while minimize lung inflammation and injury associated with mechanical ventilation (2). Avoidance of intubation and increased use of NCPAP to treat respiratory distress syndrome has been shown to decrease the incidence of chronic lung disease (3,4). However, NCPAP does have some common clinical limitations. First, the administration of NCPAP has inherent mechanical difficulties in appropriately maintaining the nasal prong apparatus within the small neonatal nose. Secondly, the nasal prongs used to deliver NCPAP can cause nasal septal trauma. Lastly, some premature infants do not tolerate the NCPAP apparatus which must be tightly affixed to their nose and face. This intolerance is often demonstrated by increased patient movement, and subsequently, the risk of mechanical difficulties and septal trauma increase during these times. Although NCPAP continues to be used in most neonatal intensive care units (NICUs), due to its aforementioned drawbacks, we continue to look for other effective, non-invasive modes of ventilation to provide support to premature infants with respiratory distress.

Humidified high flow nasal cannula (HFNC) has recently been introduced into neonatal respiratory care as a means of providing positive distending pressure to the neonate with respiratory distress. HFNC aims to maximize patient tolerance by employing heated, humidified gas flow through the standard neonatal nasal cannula that is used routinely in neonatal intensive care units. HFNC provides positive distending pressure by using high gas flow (>1 liter per minute) (5). Although numerous neonatal intensive care units are using HFNC, including both NICUs at Children's Hospitals of Minnesota, there are very few studies regarding its use in this population. Anecdotally, the premature babies tolerate the administration of HFNC quite well. However, like any new therapy, there are many unknowns.

There is only one study to date which investigates HFNC versus NCPAP in the preterm neonate (6). Sreenan and colleagues found HFNC to be as effective as NCPAP in the management of apnea of prematurity and also demonstrated that the positive distending pressure provided by HFNC varied with the patient's weight. Sreenan's study as well as preliminary data presented in abstract form cite HFNC use with various amounts of gas flow, ranging from 1 liter per minute up to 6 liters per minute (6,7,8). The choice of how much gas flow to use with the HFNC system is unclear. This decision is actually a three-fold question: 1) the initial amount of liter flow to use, 2) what does a particular liter flow provide for positive distending pressure to that patient, and 3) are these values system-specific? We aim to evaluate these questions in our study. Until recently, NCPAP has been the mainstay of non-invasive ventilatory support for premature babies. However, as HFNC is better tolerated and uses a nasal cannula that is less prone to mechanical mishaps than NCPAP, it is clear that we need more information to accurately treat babies with HFNC. The results of this study will help guide the use of HFNC in preterm babies with respiratory insufficiency, as knowledge of the positive distending pressures derived from the HFNC system are crucial in minimizing barotrauma to the fragile, premature lung.

ELIGIBILITY:
Inclusion Criteria:

* 1) receiving NCPAP ventilatory support at > 72 hrs. of age and 2) requiring FiO2 21-50% on NCPAP.

Exclusion Criteria:

* FiO2 >50%, presence of pneumothorax or pleural effusion, anatomical abnormalities of the airway, lungs, or esophagus, or cyanotic congenital heart defect.

Min Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-07; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Mean esophageal pressure | 3.5 hours

SECONDARY OUTCOMES:
Vital signs | 3.5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Mammel, MD, Principal Investigator — Children's Hospital and Clinics of Minnesota
Locations (1):
- Children's Hospital and Clinics of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Fanaroff & Martin, Ch. 42, pg.1003
- [Background] Jobe AH, Kramer BW, Moss TJ, Newnham JP, Ikegami M. Decreased indicators of lung injury with continuous positive expiratory pressure in preterm lambs. Pediatr Res. 2002 Sep;52(3):387-92. doi: 10.1203/00006450-200209000-00014. PMID 12193673
- [Background] Lindner W, Vossbeck S, Hummler H, Pohlandt F. Delivery room management of extremely low birth weight infants: spontaneous breathing or intubation? Pediatrics. 1999 May;103(5 Pt 1):961-7. doi: 10.1542/peds.103.5.961. PMID 10224173
- [Background] Gittermann MK, Fusch C, Gittermann AR, Regazzoni BM, Moessinger AC. Early nasal continuous positive airway pressure treatment reduces the need for intubation in very low birth weight infants. Eur J Pediatr. 1997 May;156(5):384-8. doi: 10.1007/s004310050620. PMID 9177982
- [Background] Locke RG, Wolfson MR, Shaffer TH, Rubenstein SD, Greenspan JS. Inadvertent administration of positive end-distending pressure during nasal cannula flow. Pediatrics. 1993 Jan;91(1):135-8. PMID 8416477
- [Background] Sreenan C, Lemke RP, Hudson-Mason A, Osiovich H. High-flow nasal cannulae in the management of apnea of prematurity: a comparison with conventional nasal continuous positive airway pressure. Pediatrics. 2001 May;107(5):1081-3. doi: 10.1542/peds.107.5.1081. PMID 11331690
- [Background] Ramanathan A, Cayabyab R, et al. High flow nasal cannula use in preterm and term newborns admitted to neonatal intensive care unit: a prospective, observational study. Pediatr Acad Soc 2005; 57:3417
- [Background] Chang GY, Cox CA, Shaffer TH. Nasal cannula, CPAP, and high-flow nasal cannula: effect of flow on temperature, humidity, pressure, and resistance. Biomed Instrum Technol. 2011 Jan-Feb;45(1):69-74. doi: 10.2345/0899-8205-45.1.69. PMID 21322815
- [Derived] Lampland AL, Plumm B, Meyers PA, Worwa CT, Mammel MC. Observational study of humidified high-flow nasal cannula compared with nasal continuous positive airway pressure. J Pediatr. 2009 Feb;154(2):177-82. doi: 10.1016/j.jpeds.2008.07.021. Epub 2008 Aug 30. PMID 18760803